CLINICAL TRIAL: NCT06213909
Title: A Retrospective Study of the Effects of Different Pathologic Phenotypes of Bullous Pemphigoid on Clinical Management and Prognosis
Brief Title: Retrospective Study of the Effects of Sub-pathologic Phenotypes of BP on Clinical Management and Prognosis
Acronym: BP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XijingH-PF-KY20232420-C-1
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-12

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- eosinophil group: Based on the histopathologic phenotype of the patient's skin, the inflammatory cells infiltrating within and around the blisters were predominantly eosinophils
  Interventions: Other: This is a retrospective analysis of health data from inpatient record, no intervention was designed
- neutrophil group: Based on the histopathologic phenotype of the patient's skin, the inflammatory cells infiltrating within and around the blisters were predominantly neutrophil
  Interventions: Other: This is a retrospective analysis of health data from inpatient record, no intervention was designed
- lymphocyte group: Based on the histopathologic phenotype of the patient's skin, the inflammatory cells infiltrating within and around the blisters were predominantly lymphocyte
  Interventions: Other: This is a retrospective analysis of health data from inpatient record, no intervention was designed

INTERVENTIONS:
Other: This is a retrospective analysis of health data from inpatient record, no intervention was designed — This is a retrospective analysis of health data from inpatient record, no intervention was designed

SUMMARY:
Bullous pemphigoid (BP) is a chronic autoimmune subepidermal blistering disease primarily affecting the elderly with a significant risk of mortality and morbidity. Various inflammatory cells such as eosinophils, lymphocytes, neutrophils and their granulopoiesis play an important role in the pathogenesis of BP. Infiltration of peripheral blood eosinophils, lymphocytes, and neutrophils into the skin is considered a major feature of BP, making it a heterogeneous disease with different histologic and clinical subtypes. This clinical study was conducted to further investigate the impact of different pathologic phenotypes of BP on the treatment and prognosis of the disease. A retrospective epidemiologic investigative approach was used，and case collection included demographic information, medical history, clinical manifestations, and histopathologic features. Including gender, age, duration of disease, number of days of hospitalization, mucosal involvement, clinical diagnosis before admission, histopathological diagnosis, laboratory tests, concomitant diseases, treatment and its changes in laboratory indexes before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients with Bullous Pemphigoid who were first hospitalized in the Department of Dermatology of Xijing Hospital
* (2) Age 0-100 years old, gender is not limited.
* (3) Diagnosis is confirmed by clinical, histopathologic, immunopathologic and/or anti-BP180 antibody tests.
* (4) Complete skin histopathology information

Exclusion Criteria:

* (1) Patients with Bullous Pemphigoid who were not first diagnosed in our hospital.
* (2) Those who have received systemic glucocorticoid, immunosuppressant, biologic, or other drug therapy within the past month.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We included patients with BP who were first admitted to the Department of Dermatology of Xijing Hospital with a clear diagnosis, complete information on skin histopathology slides, and were of any gender and age.
Sampling Method: Non-Probability Sample
Enrollment: 318 (Estimated)
Dates: Start 2024-01-11 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Bullous Pemphigoid Disease Area Index (BPDAI) severity score | 10 years
  We use BPDAI severity score as measure tool

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Phd, Principal Investigator — Dermatology Department of Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol